CLINICAL TRIAL: NCT06349421
Title: Exploring the Impact of Fully Guided Implant Placement on Classifying Bone Quality Through Tactile Sensation
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401078RINE
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Dentistry; Education
Keywords: dental implant; bone quality; tactile sensation; fully guided surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bone quality stands as a crucial determinant impacting the success rate of dental implants, exerting influence on both implant primary stability and the efficacy of osseointegration. While radiographic images can partially reveal bone quality, experienced surgeons often rely on tactile sensation during bone drilling to assess it. Subsequently, based on the diagnosed bone quality, distinct implant designs and surgical protocols have been invented to enhance survival rates.

Technological advancements now enable the preoperative design of implant placement through a comprehensive guide, merging CBCT DICOM files with digital oral scanning data. This "fully guided" approach enhances the precision, stability, and safety of implant placement surgery. However, the use of a fully guided surgical guide introduces an additional factor-the friction between the drill and guide-potentially impacting the surgeon's tactile feedback.

This study aims to assess the difference in bone quality evaluation by tactile sensation between freehand drilling and drilling with a fully guided surgical guide, using test blocks of different bone density. The discussion will explore the pros and cons of employing a fully guided guide to optimize outcomes in implant treatment.

DETAILED DESCRIPTION:
The pilot study involves five subjects, while the main experiment will include thirty subjects. The experiment consists of two rounds, each with seven simulated bone samples. These samples include four different densities (5pcf, 5pcf, 10pcf, 10pcf, 15pcf, 15pcf, 30pcf) tested in random order. Before each round of testing, participants drill into a 50 pcf bone sample and identifying it as the hardest scale. The experiment then commences with the first round employing conventional drilling tests, followed by the second round drilling with a fully guided surgical template. After each drilling session, participants assess the hardness by recording a VAS score on a 10cm scale. The evaluation criteria utilize VAS scores as the measurement tool. The aim of this experiment is to investigate whether there are differences in the classification of bone density judged by using a fully guided surgical template compared to judgments made without using the template, under the same bone density conditions. Additionally, the study aims to determine if the use of the template affects the accuracy of bone density assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified dentist
2. Practice within 10 years
3. Experience of Implant surgery should be less than 10 implants
4. Age: 24-40 y

Exclusion Criteria:

1. Unable to follow the entire test

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Board-certified dentist with age over 24 to 40 years old who has practice within 10 years and experience of Implant surgery should be less than 10 implants
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
VAS scale at the same density of sawbone | From admission to discharge, up to 1 year
  To compare the VAS scale at the same density of sawbone between free-hand drilling and drilling with fully guided stent.

CONTACTS AND LOCATIONS:
Overall Officials: wang tongmei, Study Chair — National Taiwan University
Locations (1):
- Taiwan National University, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No
The study participants only sign for this study. The personal data is promised to them should be private.